CLINICAL TRIAL: NCT03679416
Title: Is There a Benefit of Whole Body Computed Tomography (WBCT) for Patients With Only High Velocity Road Traffic Collision (RTC) Vittel Criteria?
Acronym: Cinescan
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC17-3082_Cinescan
Record Dates: First submitted 2018-09-19; First posted 2018-09-20 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: High Velocity Transport Accidents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
For victims of high velocity RTC, with no other Vittel criteria of gravity, normal clinical examination of the thorax, abdomen and pelvis and Glasgow Coma Scale (GCS) score of 15 :

* Study of clinically unsuspected injuries discovered on WBCT
* Description
* Predictive factors
* Diagnostic performances of kinetic elements of Vittel criteria, and results of examinations realised at the ED.

ELIGIBILITY:
Inclusion Criteria:

Consecutives patients consulting the emergency department between August 1st 2016 and July 31th 2017 :

* Older than 18 y.o.
* WBCT performed,
* Victim of a high velocity RTC as defined by the presence of at least one criteria of the kinetics elements of the Vittel Criteria
* Normal physical exam of the chest, abdomen and pelvis,
* GCS score of 15

Exclusion Criteria:

* Opposition of the patient to the use of their CT-scan for research
* Patients who are under legal protection
* Patients who are incarcerated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: victims of high velocity RTC, with no other Vittel criteria of gravity, normal clinical examination of the thorax, abdomen and pelvis and Glasgow Coma Scale (GCS) score of 15.
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Number of injuries diagnosed by Whole Body Computed Tomography (WBCT) that were not clinically suspected. | The day of inclusion
  Number of injuries diagnosed by WBCT that were not clinically suspected.
  Classification in 3 categories according to their management :
  * Potentially severe, that involve modification of patients management
  * Injuries that could require further investigation according to the symptoms
  * Minor injuries that require no further investigation or specific management

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Rennes, Rennes, France